CLINICAL TRIAL: NCT06177535
Title: The Effect of Oral Kavalactones on Cortisol, Measures of Burnout, and Motivation in Nurses
Brief Title: A Study of Oral Kavalactones Effect on Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-005268
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Stress
Keywords: Nursing Professionals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kava Group (Experimental): Subjects will receive Kavalactones for 28 days
  Interventions: Dietary Supplement: Kavalactones
- Placebo Group (Placebo Comparator): Subjects will receive placebo for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Kavalactones — Three 75 mg capsules orally once daily within one hour of bedtime (225 mg total/day)
  Arms: Kava Group
Drug: Placebo — Three capsules orally once daily within one hour of bedtime. Looks exactly like the study drug, but it contains no active ingredient.
  Arms: Placebo Group

SUMMARY:
This research study is being done to assess the impact of taking Kava extract (Piper methysticum), a dietary supplement on cortisol in a healthy nursing population.

ELIGIBILITY:
Inclusion Criteria:

* Surgical services nurses at Mayo Clinic in Rochester, MN.
* Able to participate fully in all aspects of the study.
* Willing to use birth control for the duration of the study (if of childbearing potential).
* Understood and signed study informed consent.

Exclusion Criteria:

* Pregnant, nursing, or trying to conceive.
* Persons with a menstrual cycle who are not willing and able to use an approved contraceptive during the study (female sterilization (tubal ligation, hysterectomy), IUD or another implant, oral or injectable contraceptive, contraceptive patch/ring, diaphragm/cervical cap, male sterilization (vasectomy), male condom, female condom, sponge/spermicide) (Persons who do not have sex with men can participate without the use of an approved contraceptive).
* Use of kava or kava-containing products within the past 8 weeks.
* Any prior adverse reaction or known sensitivity or allergy to kava or related botanicals (peppers).
* Use of acetaminophen that cannot be discontinued or replaced with an NSAID during the study.
* Use of oral corticosteroids (e.g., hydrocortisone) or other steroids (e.g., prednisone).
* Alcohol use greater than 1 drink per day.
* Use of kratom within the past 8 weeks.
* Recent history of clinical depression or anxiety diagnosis.
* Known significant liver disease or dysfunction.
* Known significant kidney disease or dysfunction.
* Known Addison's or Cushing's Disease.
* Known catecholamine imbalance or medication use which influences catecholamine levels.
* History or current diagnosis of cancer (except for successfully treated basal cell carcinoma diagnosed less than 5 years prior to screening or cancer in full remission more than 5 years after diagnosis).
* Recent history or acute disease or unstable medical condition.
* Surgery planned during the course of the trial.
* A known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Cortisol | Baseline, 4 weeks
  Blood serum cortisol levels reported in micrograms per deciliter (mcg/dL)

SECONDARY OUTCOMES:
Change in burnout | Baseline, 4 weeks
  Measured using the Maslach Burnout Inventory-Human Services Survey for Medical Personnel - MBI-HSS (MP): The MBI-HSS (MP) addresses three scales: Emotional Exhaustion measures feelings of being emotionally overextended and exhausted by one's work; Depersonalization measures an unfeeling and impersonal response toward patients; Personal Accomplishment measures feelings of competence and successful achievement in one's work.
Change in motivation | Baseline, 4 weeks
  Measured using the Cravings for Rest and Volitional Energy Expenditure (CRAVE) survey developed to measure motivation states for physical activity and sedentary behaviors. Subjects indicate how much they want or desire to perform activities by circling the number along each line between 0 (not at all) and 10 (more than ever).
Change in mood | Baseline, 4 weeks
  Measured using the Depression, Anxiety and Stress Scale - 21 Items (DASS-21). The DASS-21 is a non-diagnostic, validated instrument to assess perceived levels of depressed, stressed, or anxious emotional states over the past seven days. Scores for each state range from 0-42 and can be summed to generate a total score reflecting overall negative mood.
Change in sleep | Baseline, 4 weeks
  Measured using the PROMIS Sleep Disturbance -Short Form 6a to assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep.
Change in quality of life | Baseline, 4 weeks
  Measured using the Linear Analogue Self-Assessment (LASA) - LASA-1 single item Likert scale of 10 points (0-10) which measures quality of life, with higher score indicating better quality of life.
Change in stress | Baseline, 4 weeks
  Measured using The Perceived Stress Scale-10 (PSS) that elicits self-reported personal stress levels. The scores range from 0-40, with higher scores indicating more severe stress.
Change in cognition | Baseline, 4 weeks
  Measured using CNS Vital Signs in-office neurocognitive testing, a non-invasive clinical procedure to efficiently and objectively assess a broad spectrum of brain function performance or domains under challenge (cognition stress test).
Adverse events | 4 weeks
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials